CLINICAL TRIAL: NCT06974864
Title: Burnout vs Resilience: A Cross-sectional Study Among Healthcare Workers After the Recent Aggression in Lebanon
Brief Title: Burnout vs Resilience Among Healthcare Workers After the Recent Aggression in Lebanon
Status: Completed | Type: Observational
Sponsor: Hopital Libanais Geitaoui (Other)
Responsible Party: Principal Investigator, Mazen El Jamal, Principal Investigator, Lebanese University
Other Study IDs: 2025-IRB-04
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Burnout; Resilience
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the extent of burnout and the prevalence of resilience traits among healthcare workers in Lebanon, specifically after the recent Israeli aggression. This study will also explore factors related to burnout and resilience, as well as the relationship between resilience and mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers currently working in Lebanon including physicians, nurses, and other allied health workers (physiotherapists, psychologists, radiology technicians, occupational therapist, midwives, paramedics…).
* Students/interns training in these professions are also included.

Exclusion Criteria:

* non-healthcare staff
* healthcare workers who stopped working during war

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Oldenburg Burnout Inventory (OLBI) scale | February 2025
  The OLBI scale contains 16 items and uses a 4-point Likert scale. Total scores range from 16 to 64. Higher scores indicated higher burnout levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese Hospital Geitaoui, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No